CLINICAL TRIAL: NCT00694018
Title: Veterans Walk to Beat Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIR 07-177
Record Dates: First submitted 2008-05-28; First posted 2008-06-10 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-09

CONDITIONS: Back Pain
Keywords: randomized trial; walking
MeSH Terms: conditions — Back Pain | interventions — Educational Status; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education and Standard Care (Active Comparator): Received standard care and participated in an educational program for individuals with chronic back pain. Also received an uploading pedometer but no feedback or goals about their walking activity.
  Interventions: Other: Education and standard care
- Internet Mediated Enhanced Pedometer (Experimental): In addition to standard care and participating in an educational program, participants received an enhanced pedometer for uploading step information, e-mail messages with weekly step goals and access to a website that provided step goals and feedback, tailored motivational messages and on on-line community for communication asynchronously with staff and other participants.
  Interventions: Other: Education and standard care; Behavioral: Internet mediated enhanced pedometer intervention

INTERVENTIONS:
Other: Education and standard care — Educational program for individuals with chronic back pain.
Behavioral: Internet mediated enhanced pedometer intervention — Enhanced pedometer for uploading step information and website that provides step goals and feedback, tailored motivational messages and an online community.
  Arms: Internet Mediated Enhanced Pedometer

SUMMARY:
The objective of this study was to assess whether an Internet-mediated pedometer based intervention would increase walking and improve function among individuals with chronic back pain.

DETAILED DESCRIPTION:
Project Background/Rationale: Chronic pain, and especially back pain, is common among VA patients, affecting approximately 60% of veterans using VA primary care services. Chronic pain is associated with increased disability, poorer health status, anxiety and depression, decreased quality of life, decreased employment and increased health services use and costs. Current evidence suggests that exercise is one of the most effective strategies for managing chronic pain. However, there are few clinical programs that use generally available tools and a relatively low cost approach to help patients with chronic back pain initiate and maintain an exercise program.

Project Objectives: The primary objective of this study was to assess the efficacy of an Internet-mediated pedometer based intervention that was designed to increase walking and improve pain-related function among individuals with chronic back pain. The Specific Aims of this randomized, controlled trial were: 1) To determine whether an internet-mediated pedometer based intervention will reduce pain-related functional interference among patients with chronic back pain in the short term and over a 12-month timeframe; 2) To assess the effect of the intervention on walking (measured by step counts), quality of life, pain intensity, pain related fear and self-efficacy for exercise among patients with chronic back pain; and 3) To identify factors associated with a sustained increase in walking over a 12-month timeframe among patients randomized to the intervention.

Project Methods: We conducted a randomized controlled trial of an Internet-mediated, pedometer based intervention to promote walking and improve pain-related function among patients with chronic back pain compared to enhanced usual care. Participants were followed for 12 months to investigate the efficacy of the intervention in assisting patients with initiating and maintaining a regular walking program and improving pain-related function. We recruited patients with chronic back pain (primarily low back pain) receiving care at one VA health care system. Study patients were randomized to one of two groups: 1) enhanced usual care or 2) the Internet-mediated, pedometer based intervention. All participants attended an educational program designed specifically for individuals with chronic back pain. Study participants randomized to the intervention were given an enhanced pedometer and access to a study website that provided step goals and feedback, tailored motivational messages and an e-community. Those in the control group received a pedometer but did not have access to the website. Both groups completed on-line survey assessments at baseline, 6, and 12 months and were asked to report adverse events on a regular basis. The primary outcome for this study was pain-related functional interference. Secondary outcomes included average daily steps at 12 months as measured using the study pedometer, health related quality of life, pain intensity, pain related fear and self-efficacy for exercise. The analysis was conducted based on intention to treat principles and used multivariable modeling procedures to determine the effect of the intervention on our outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving care at the VA Ann Arbor Healthcare System
* Have back pain that has persisted for more than 3 months
* Have a sedentary lifestyle (less than 150 minutes of physical activity per week)
* Have access to a computer (with Windows XP or Vista) on at least a weekly basis with an available USB port and Internet access
* Have a working e-mail address
* Are competent to provide written informed consent
* Are able to communicate in English
* Are not institutionalized
* Can identify a health care provider who can provide medical clearance.

Exclusion Criteria:

* Currently pregnant
* Cannot walk at least one block
* Cannot obtain written clearance to start a walking program from a treating healthcare provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2009-05; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L. Krein, PhD RN, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Krein SL, Kadri R, Hughes M, Kerr EA, Piette JD, Holleman R, Kim HM, Richardson CR. Pedometer-based internet-mediated intervention for adults with chronic low back pain: randomized controlled trial. J Med Internet Res. 2013 Aug 19;15(8):e181. doi: 10.2196/jmir.2605. PMID 23969029
- [Result] Krein SL, Metreger T, Kadri R, Hughes M, Kerr EA, Piette JD, Kim HM, Richardson CR. Veterans walk to beat back pain: study rationale, design and protocol of a randomized trial of a pedometer-based internet mediated intervention for patients with chronic low back pain. BMC Musculoskelet Disord. 2010 Sep 13;11:205. doi: 10.1186/1471-2474-11-205. PMID 20836856
- [Derived] Krein SL, Bohnert A, Kim HM, Harris ME, Richardson CR. Opioid use and walking among patients with chronic low back pain. J Rehabil Res Dev. 2016;53(1):107-16. doi: 10.1682/JRRD.2014.08.0190. PMID 26934620

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education and Standard Care | Internet Mediated Enhanced Pedometer
Started | 118 | 111
6 Months | 106 | 101
Completed | 105 | 102
Not Completed | 13 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education and Standard Care | Internet Mediated Enhanced Pedometer | Total
Number analyzed (Participants) | 118 | 111 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.8) | 51.2 (12.5) | 51.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 102 | 99 | 201
Race/Ethnicity, Customized [Number; unit: participants]
  White | 101 | 82 | 183
  Black | 11 | 14 | 25
  Other or prefer not to answer | 6 | 15 | 21
Region of Enrollment [Number; unit: participants]
  United States | 118 | 111 | 229
Roland Morris Disability Questionnaire (RDQ) Score [Mean (Standard Deviation); unit: units on a scale] — The Roland Morris Disability Questionnaire score ranges from 0-24, with higher scores indicating greater disability.
  units on a scale | 9.8 (5.7) | 9.1 (6.0) | 9.5 (5.8)
Daily step counts [Mean (Standard Deviation); unit: steps] | 4321.9 (2285.4) | 4492.9 (2749.9) | 4404.8 (2517.0)

OUTCOME MEASURES:

1. Primary Outcome: The Roland Morris Disability Questionnaire (RDQ) Score
Description: The Roland Morris Disability Questionnaire score ranges from 0 to 24, with higher scores indicating greater disability
Time Frame: 12 months
Population: The number of participants analyzed is slightly lower than the number who completed the study at 12 months due to item non-response on the final study survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education and Standard Care | Internet Mediated Enhanced Pedometer
Number analyzed (Participants) | 103 | 102
units on a scale | 8.3 (5.6) | 6.6 (5.9)

ADVERSE EVENTS:
Time Frame: During the 1 year intervention period
Description: Participants reported any health problems whether or not study related as prompted by weekly (intervention) or monthly (control) emails. After the first four weeks and then every eight weeks after that, all participants were prompted to complete a survey on the website that asked about specific adverse events and symptoms.
Arm/Group | Education and Standard Care | Internet Mediated Enhanced Pedometer
Serious Adverse Events (participants affected / at risk) | 26/118 | 27/111
Other Adverse Events (participants affected / at risk) | 76/118 | 87/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Education and Standard Care (N=118) | Internet Mediated Enhanced Pedometer (N=111)
All serious adverse events (General disorders) | 26 | 27 — serious adverse events during the study period ranged from hospitalizations for planned surgeries to death. All were reviewed and none were found to be study-related. They were reported but not categorized by system.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Education and Standard Care (N=118) | Internet Mediated Enhanced Pedometer (N=111)
All (non-serious) adverse events (General disorders) | 76 | 87 — We have overall events/person/group but only number of events by system/group. The most common events: worsening back pain (74 education, 85 pedometer), musculoskeletal (36 education, 76 pedometer) and cardiovascular (37 education, 48 pedometer)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes